CLINICAL TRIAL: NCT02557074
Title: TREg Activation in the Treatment of the PELADE (Alopecia Areata). Double Blind Randomized Placebo Controlled Comparative Study Using Low Doses of IL2
Brief Title: TREg Activation in the Treatment of the PELADE (Alopecia Areata)
Acronym: TreatPelade
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-API-01
Record Dates: First submitted 2015-08-11; First posted 2015-09-22 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IL2 - Group A (Experimental): Patient will received IL2 low doses (1.5 to 3MUI/d) -
  * IL2 1.5MUI/d SC from day 1 to day 5 for the first course of treatment
  * IL2 3MUI/d SC from day 1 to day 5 for the 3 following courses
  Interventions: Drug: IL2
- Placebo - Group B (Placebo Comparator): NaCl 9% serum (placebo) NaCl 9% serum SC from day 1 to day 5 for the four courses of treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IL2 — IL2 1.5MUI/d SC from day 1 to day 5 for the first course of treatment IL2 3MUI/d SC from day 1 to day 5 for the 3 following courses
  Arms: IL2 - Group A
Drug: placebo — NaCl 9% serum SC from day 1 to day 5 for the four courses of treatment
  Arms: Placebo - Group B

SUMMARY:
In a prospective pilot study the investigators showed that low doses of IL2 could be beneficial for severe AA inducing a long lasting regrowth in 4 out of the 5 patients treated.

The objective of this study is to compare the long term efficacy of low doses of IL2 versus placebo in a multicenter prospective randomized double blind study.

ELIGIBILITY:
Inclusion Criteria:

* Of more than 18 years old,
* Affiliated to the social security system,
* Clinical diagnosis of alopecia areata,
* 50 % of the surface of the scalp affected
* Last flaire started less than one year
* Alopecia areata resisting to at least 1 systematic treatment including phototherapy (UVB or PUVA), general corticosteroid therapy or methotrexate
* Signature of the informed consent

Exclusion Criteria:

* Pregnancy or refusal of contraception at the women old enough to procreate,
* Refusal of contraception at the men
* Local treatment (dermocorticoïdes, minoxidil) or systematism (oral corticosteroid therapy, méthotrexate or the other immunosuppresseur) since less than 2 less,
* Evolutionary autoimmune cancer or disease or in forgiveness
* Excessive grip(taking) of alcohol (upper to 3 glasses of wine a day or one pre-lunch drink a day)
* Seropositivity VHC, VHB, or HIV
* Patient presenting a severe renal and/or hepatic insufficiency,
* Presenting patient one zoned, the chicken pox, the herpes, the tuberculosis, an evolutionary infectious disease, a respiratory failure …
* Vulnerable person (nobody under guardianship minor(miner), adults, deprived of freedom)
* IC in the treatment(processing) by IL-2R
* Presenting a contraindication to ProleukinR

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Score Salt | Once : at 12 months post-treatment
  Success defined by a SALT score lower or equal to 25 at the end the study (12 months post-treatment). It will be calculated by 2 physicians blinded to the treatment received on standardized pictures.

SECONDARY OUTCOMES:
Quality of life | at one day, 22 days, 43 days, 64 days, 251 days, 434 days
  The quality of life (QdV) will be estimated with the scale DLQI which is a scale of QdV validated for the dermatological diseases.
Adverse Event | at one day, 22 days, 43 days, 64 days, 251 days, 434 days
  The tolerance will be clinically and biologically estimated at each visit. The type and the rank of every AE will be raised.
Satisfaction of patient | at 12 months post-treatment
  The satisfaction of the patients will be estimated on an analog visual scale(ladder) going of 0 (not satisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PUPH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (6):
- France (6):
  - AP-HM - La timone - Dermatologie, Marseille, Bouche Du Rhône
  - CHU de Nimes - Dermatologie, Nîmes, Languedoc-Roussillon
  - CHI St Raphael Fréjus - Dermatologie, Fréjus, PACA
  - CHU Montpellier - Dermatologie, Montpellier
  - CHU de Nice - dermatologie, Nice
  - AP-HP St Louis - Dermatologie, Paris, Île-de-France Region